CLINICAL TRIAL: NCT00992134
Title: Immunochemotherapy With Rituximab-Bendamustine-Cytarabine for Patients With Mantle Cell Lymphoma Not Eligible for Intensive Regimens or Autologous Transplantation.
Brief Title: Immunochemotherapy With Rituximab-Bendamustine-Cytarabine (R-BAC) for Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Bortolo Hospital (Other)
Responsible Party: Principal Investigator, Carlo Visco, MD, St. Bortolo Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI-1903; EudraCT 2009-009912-34
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2010-09

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Lymphoma, Mantle-Cell; Bendamustine; Cytarabine; Rituximab; Treatment; Combination chemotherapy
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Bendamustine Hydrochloride; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab, Bendamustine, Cytarabine — Rituximab IV 375 mg/m2 on day 1. Bendamustine IV 70 mg/m2 over a 30-60 minute infusion on day 1 and 2. Cytarabine IV 800 mg/m2, over a 2-hour infusion, 2 hours after Bendamustine, on Day 1, 2, and 3.
  Four to six cycles. Recycle every 28 days.
  Other Names: Ribomustin; Mabthera; Ara-C

SUMMARY:
The objective of the study is to demonstrate the safety, tolerability, and activity of Rituximab-Bendamustine-Cytarabine(R-BAC) regimen in patients with mantle cell lymphoma (MCL) aged 65 years or more, as well as in younger patients who are not eligible for intensive regimens including/not including autologous transplantation.

DETAILED DESCRIPTION:
Since Bendamustine has recently shown promising safety and efficacy in combination with monoclonal antibodies in the treatment of patients with MCL, the goal of this study is to investigate the possible therapeutic benefit of combining Ara-C with Bendamustine and Rituximab (R-BAC). All three agents exhibit individual and unique mechanisms of action in MCL, and a synergistic or additive effect might be expected when these agents are used in combination, as suggested by the pre-clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with MCL aged 65 years or more, or <65 years if not eligible for intensive treatments including/not including autologous transplantation.
* MCL patients of any age who relapse/progress or are resistant after one line of chemotherapy.
* CD20+ .
* Karnofsky score of at least 70%
* Adequate renal function (Creatinine clearance >40 mL/min), with preserved diuresis.
* Adequate liver function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) <2.5 x upper limit of normal (ULN) value, total bilirubin <2 mg/dL, unless directly attributable to the patient's tumor.
* Negative serum pregnancy test 1 week prior to treatment both for pre-menopausal women and for women who are <2 years after onset of menopause.
* Hepatitis B core antibody (HBcAb) positive patients may be enrolled if correct antiviral prophylaxis is administered at least 2 weeks before initiating protocol treatment.
* Written informed consent.

Exclusion Criteria:

* Prior treatment with Bendamustine.
* Refractoriness to Rituximab, defined as progressive disease during a previous cycle including this drug, or relapse within 6 months to any previous cycle including Rituximab.
* Previous Rituximab infusion-related severe reactions.
* Human immunodeficiency virus (HIV) positive.
* Medical conditions or organ injuries that could interfere with administration of therapy.
* Active bacterial, viral, or fungal infection requiring systemic therapy.
* Seizure disorders requiring anticonvulsant therapy.
* Severe chronic obstructive pulmonary disease with hypoxaemia.
* History of severe cardiac disease: New York Heart Association (NYHA) functional class III-IV, myocardial infarction within 6 months, ventricular tachyarrhythmias, dilatative cardiomyopathy, or unstable angina.
* Uncontrolled diabetes mellitus.
* Active secondary malignancy.
* Known hypersensitivity or anaphylactic reactions to murine antibodies and proteins (for patients treated with Rituximab), to Bendamustine or mannitol.
* Fertile men and women of childbearing potential unless surgically sterile or using adequate measures of contraception.
* Major surgery within 4 weeks of study Day 1.
* HBsAg+ and HCV+ patients
* Any co-existing medical or psychological condition that would preclude participation in the study or compromise the patient's ability to give informed consent, or that may affect the interpretation of the results, or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of R-BAC treatment will be tested to determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of Ara-C when combined with Bendamustine and Rituximab. | June 2011

SECONDARY OUTCOMES:
Overall response and freedom from progression after R-BAC treatment | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Visco, MD, Principal Investigator — Department of Hematology, San Bortolo Hospital, Vicenza
Locations (1):
- Department of Hematology, Ospedale San Bortolo, Vicenza, VI, Italy

REFERENCES:
- [Derived] Visco C, Finotto S, Zambello R, Paolini R, Menin A, Zanotti R, Zaja F, Semenzato G, Pizzolo G, D'Amore ES, Rodeghiero F. Combination of rituximab, bendamustine, and cytarabine for patients with mantle-cell non-Hodgkin lymphoma ineligible for intensive regimens or autologous transplantation. J Clin Oncol. 2013 Apr 10;31(11):1442-9. doi: 10.1200/JCO.2012.45.9842. Epub 2013 Feb 11. PMID 23401442